CLINICAL TRIAL: NCT01456338
Title: Cognitive Behavioral Therapy for PTSD in Addiction Treatment: A Randomized Pilot Trial
Brief Title: Cognitive Behavioral Therapy for Post Traumatic Stress Disorder in Addiction Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mark McGovern, Associate Professor of Psychiatry and of Community and Family Medicine, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5K23DA016574_PILOT; 5K23DA016574 (NIH)
Record Dates: First submitted 2011-10-03; First posted 2011-10-20 (Estimated); Last update posted 2011-10-20 (Estimated); Status verified 2011-10

CONDITIONS: Stress Disorders, Post-Traumatic; Substance-Related Disorders
Keywords: cognitive behavior therapy; addiction; posttraumatic stress disorder (PTSD)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders; Behavior, Addictive | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral Therapy (Experimental): Cognitive Behavioral Therapy (CBT) is a non-exposure based, manual-guided individual therapy. CBT for PTSD consists of 3 learning and skill components designed to improve PTSD symptoms and substance use: 1) Patient education about PTSD and its relation to substance use and treatment; 2) Breathing retraining: A behavioral anxiety reduction skill; and 3) Cognitive restructuring: A cognitive approach and functional analysis of the link among emotions, cognitions and situations.
  Interventions: Behavioral: Cognitive Behavioral Therapy for PTSD
- Individual Addiction Counseling (Active Comparator): Individual Addiction Counseling (IAC) was adapted from the Individual Drug Counseling (IDC) manual used in the NIDA Cocaine Collaborative Study. IAC is a manual-guided treatment that focuses on substance use and history of use, consequences of use and denial, developing strategies for relapse prevention, and facilitation of connection with peer recovery support groups, specifically twelve step groups. The current adaptation of IAC modified the IDC manual by broadening the focus to include drugs other than cocaine, as well as alcohol.
  Interventions: Behavioral: Individual Addiction Counseling

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for PTSD — Individual CBT, approx. 12 sessions, one session per week
  Other Names: CBT for PTSD; CBT
  Arms: Cognitive Behavioral Therapy
Behavioral: Individual Addiction Counseling — Individual therapy, approx. 12 sessions, one session per week
  Other Names: IAC
  Arms: Individual Addiction Counseling

SUMMARY:
The purpose of this phase of the study is to further assess the efficacy of cognitive behavioral therapy (CBT) for posttraumatic stress disorder (PTSD), as delivered by routine addiction counselors, and to compare CBT for PTSD with individual addiction counseling (IAC) on our primary outcomes.

DETAILED DESCRIPTION:
The main hypothesis being tested is that a cognitive behavioral therapy (CBT) for posttraumatic stress disorder (PTSD) can improve treatment retention and outcomes for both posttraumatic stress and substance use disorders. The investigators have completed a Safety & Practicality Study and a Feasibility Study and both studies found that CBT for PTSD was safe and effective in reducing PTSD symptoms, improving retention, and in reducing substance use. The present study proposes to continue testing the hypotheses by evaluating and comparing the PTSD, retention and substance use outcomes resulting from CBT versus a control condition. This is termed the "Pilot Trial" phase of behavioral therapy development and requires comparing the investigational treatment (CBT) with a control treatment, within the context of addiction treatment-as-usual (intensive outpatient programs or methadone maintenance clinic settings). The results of this study will then be used to develop a RO1 grant application to NIDA to support a Stage II efficacy study (randomized controlled trial).

Our objective is to test the following specific hypotheses:

CBT for PTSD (plus addiction treatment-as-usual) vs. IAC (plus addiction treatment-as-usual): 1) Reduces PTSD symptoms; 2) Improves addiction treatment retention; and, 3) Reduces substance use and severity. A hierarchy of effects is hypothesized. The target of the CBT is PTSD symptoms, which if reduced, will favorably leverage both treatment retention and substance use, above and beyond the equivalence in type and amount of treatment in both conditions.

This study involves is a two-group repeated measures design. Within the NIDA stage model, it is a randomized, pilot trial with a matched-attention control condition. The investigators plan to examine outcomes associated with the intervention versus control condition among patients receiving outpatient addiction treatment services (intensive outpatient program or methadone maintenance program). The investigators will employ assessments at baseline, during therapy, post-therapy, and three-month follow-up. Eligible subjects will be randomly assigned to the study CBT therapy (plus addiction treatment-as-usual) or the matched attention control condition (individual addiction counseling [IAC] plus addiction treatment-as-usual), and all will be followed for the research assessments regardless of whether they drop out of treatment early (whenever possible).

Patients admitted to the participating addiction treatment programs are routinely screened for PTSD using a brief self-report survey, the PTSD Checklist (PCL). These forms are collected by clinical staff of the treatment program and scored for PTSD diagnostic criteria. Patients scoring 44 or greater on the PCL are approached by a clinic staff about potential interest in the study. If they wish to learn more about the study, the research coordinator (an on-site employee) is contacted, a suitable time arranged, and the patient engaged in the process of informed consent.

If consent is granted, the subject completes the baseline assessment. The baseline assessment consists of measures gathered via interview by a member of the research team, self-administered surveys completed directly by the subject, and review of the subject's medical record to extract demographic, substance use, and treatment history information, as well as chart diagnoses.

The interview portion of the assessment consists of:

* Standardized interviews designed to assess PTSD and borderline personality disorder, another commonly associated psychiatric disorder: Clinician Administered PTSD Scale (CAPS) and the SCID-Axis II borderline personality disorder.
* A urine screen and breathalyzer to test for alcohol and other drugs.
* Standardized follow-back method for gathering data on recent alcohol and drug use: Time-line Follow-back Calendar (TLFB).

The self-administered portion of the assessment consists of measures designed to assess:

* Depression (Beck Depression Inventory-II [BDI-II])
* Anxiety (Beck Anxiety Inventory [BAI])
* Alcohol and drug use, as well as associated problems in other life areas such as medical, employment, legal, social, and psychiatric (Addiction Severity Index [ASI])
* Level of risk for HIV (HIV-risk Screening Instrument [HSI])
* Treatment utilization (Recent Treatment Survey).

If the subject continues to meet criteria for PTSD (i.e., the CAPS interview confirms diagnosis of DSM-IV PTSD, with symptom severity at 44 or higher), he or she is randomized to receive the study CBT therapy or the control condition (IAC).

At monthly (every four weeks) intervals during the provision of CBT or IAC, the subject will complete the RTS and a trauma event checklist based on the PCL, and will be tested for alcohol use (breathalyzer) and drug use (urine screen). The subject will also complete the Working Alliance Inventory (WAI - client version) at the first monthly assessment only.

Upon completion of the CBT or IAC, a member of the research team will re-interview the subject. The post-therapy assessment (approx. 3-months post-baseline) will consist of the same measures administered at baseline, with the exception of the borderline personality disorder interview.

The final research assessment is conducted three months after the post-therapy assessment. This assessment will consist of the same measures used at the post-therapy assessment, along with the trauma event checklist (to assess for re-traumatization).

The investigators plan to enroll approximately 100 subjects in the study. Based on our previous data, the investigators expect that 60% of referred subjects will actually meet eligibility criteria, leaving 60 subjects to be randomized (30 to CBT and 30 to IAC). The subject outcome and program experiences with the protocol will be used in planning the subsequent federal grant application for a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old;
2. Actively enrolled in outpatient addiction services and meets criteria for any substance use disorder;
3. Screened positive for PTSD (results of PCL show a likely Criterion A Traumatic event and a score equal to or greater than 44);
4. Willing and able to provide informed consent to participate in the study;
5. Diagnosis of PTSD verified by the CAPS and total symptom score equal to or greater than 44;

Exclusion Criteria:

1. Acute psychotic symptoms (however, persons with a psychotic disorder are eligible if their symptoms are stable and they are well-connected with appropriate mental health services);
2. Psychiatric hospitalization or suicide attempt in the past month (however, if the hospitalization or attempt was directly related to substance intoxication or detoxification and the person is currently stable, they are eligible);
3. Medical and legal situations are unstable such that ability to participate in the full duration of the study seems unlikely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2007-06; Primary Completion 2009-04 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Decrease from baseline in Clinician Administered PTSD Scale (CAPS) score (PTSD symptom severity) at 3-months and at 6-months | Baseline, 3-month, & 6-month follow-up

SECONDARY OUTCOMES:
Difference in treatment retention between ICBT and IAC at treatment completion, approx. 12 weeks | From date of treatment commensement until treatment completion, assessed up to 12 weeks
Reduction from baseline in substance use severity (Addiction Severity Index [ASI]) at 3-months and at 6-months | Baseline, 3-month & 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Mark P. McGovern, Ph.D., Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (6):
- United States (6):
  - Hartford Dispensary, Hartford, Connecticut
  - Addiction Treatment Program at DHMC, Lebanon, New Hampshire
  - Farnum Center, Manchester, New Hampshire
  - WestBridge, Manchester, New Hampshire
  - Starting Now - Brattleboro Retreat, Brattleboro, Vermont
  - Quitting Time - Clara Martin Center, Wilder, Vermont